CLINICAL TRIAL: NCT04169035
Title: The BD Odon DeviceTM for Assisted Vaginal Birth: a Feasibility Study to Investigate Safety and Efficacy
Acronym: ASSIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P/2019/435
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Pregnant Woman
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Odon device (Experimental): The practitioner providing the woman's care in labour determines that she requires an assisted vaginal birth, and there is no obstetric indication for an alternative method of assiste vaginal birth. Odon trained practitioner available to assist the birth.
  Interventions: Device: The BD Odon DeviceTM is a new device for AVB that has been designed by a team of midwives, doctors and engineers.
- Forceps or ventouse (Active Comparator): The practitioner providing the woman's care in labour determines that she requires an assisted vaginal birth, and there is no obstetric indication for an alternative method of assisted vaginal birth.
  The woman is unable to have an Odon assisted birth as no Odon trained practitioner is available to assist the birth.
  Interventions: Procedure: forceps or ventouse

INTERVENTIONS:
Device: The BD Odon DeviceTM is a new device for AVB that has been designed by a team of midwives, doctors and engineers. — The BD Odon DeviceTM works by placing a cuff of air attached to a plastic sleeve, around the baby's head. The doctor then gently pulls on this sleeve and air cuff to assist the birth of the baby.
  Arms: Odon device
Procedure: forceps or ventouse — The woman is unable to have an Odon assisted birth as no Odon trained practitioner is available to assist the birth.
  Forceps is a metal instrument with two handles used to encircle a baby's head and assist in birth.
  Ventouse is a device used to help a baby be born by putting it over the baby's head and using suction (= removing air) to pull the baby out of the mother's body.
  Arms: Forceps or ventouse

SUMMARY:
Besancon ASSIST study will investigate if the BD Odon DeviceTM is safe, effective and acceptable to women and maternity staff for assisted vaginal birth.

ELIGIBILITY:
Inclusion Criteria:

* The woman is ≥18 years of age
* The woman has a singleton pregnancy
* The pregnancy is ≥28+0 weeks' gestation
* There is a negative antenatal screen for HIV and Hepatitis B

Exclusion Criteria:

* The woman does not fulfil all of the inclusion criteria listed
* There is a diagnosis of a fetal skull abnormality precluding AVB (i.e. macrocephaly)
* There is a known osteogenesis imperfecta affected pregnancy
* There is suspicion of a fetal bleeding disorder (von Willebrand's disease, AITP, haemophilia)
* There is an intrauterine fetal death in the current pregnancy
* The woman is sensitive to latex
* The woman is currently serving a prison sentence
* The woman lacks capacity to consent
* The woman has a lack of ability to read or understand French as this would preclude successful completion of questionnaires
* The woman has received intramuscular or intravenous opiates (i.e. pethidine or morphine) within the past 6 hours
* The woman is in established labour (≥ 4cm cervical dilatation) without regional analgesia in place

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 104 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Rate of births successfully assisted with the BD Odon Device | 3 months after delivery
  Successful vaginal birth with the BD ODON DeviceTM: successful BD Odon assisted birth in the absence of maternal and neonatal serious adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mottet N, Hotton E, Eckman-Lacroix A, Bourtembourg A, Metz JP, Cot S, Poitrey E, Delhomme L, Languerrand E, Nallet C, Lallemant M, Draycott T, Riethmuller D. Safety and efficacy of the OdonAssist inflatable device for assisted vaginal birth: the BESANCON ASSIST study. Am J Obstet Gynecol. 2024 Mar;230(3S):S947-S958. doi: 10.1016/j.ajog.2023.05.016. Epub 2023 Aug 1. PMID 38462265